CLINICAL TRIAL: NCT06811402
Title: Combinaison of Virtual Reality and Rehabilitation to Improve Muscle Function, Exercise Tolerance, Exertional Symptoms and Dyspnea in Patients with Chronic Respiratory Disease: a Randomized Cross-over Trial
Acronym: OVERMUSCLED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: OVERMUSCLED
Record Dates: First submitted 2025-01-30; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Patient will undergo the rehabilitation session as the usual without the virtual reality mask.
- VR (Experimental): the patient will undergo the rehabilitation session with a virtual reality mask
  Interventions: Other: virtual reality

INTERVENTIONS:
Other: virtual reality — the patient will wear a VR mask during the session
  Arms: VR

SUMMARY:
Chronic respiratory diseases, such as Chronic Obstructive Pulmonary Disease (COPD), are a leading cause of death globally. These diseases not only contribute significantly to mortality but also lead to a decline in physical capacity, limiting daily activities and perpetuating a vicious cycle of deconditioning. Dyspnea (shortness of breath) is a major symptom, seen in 56 to 98% of COPD patients, and is linked to decreased exercise tolerance and muscle dysfunction. It often leads to reduced physical activity, further worsening respiratory function and quality of life. Dyspnea severity is associated with increased mortality, hospitalizations, and anxiety. The main therapeutic approach for these patients is pulmonary rehabilitation, which improves exercise tolerance, quality of life, and reduces hospitalizations and exacerbations. However, dyspnea limits exercise and is often a barrier to continued physical activity.

Virtual reality (VR) technology has shown promise in managing symptoms like pain, anxiety, and dyspnea by providing a distraction. Studies suggest that VR can improve dyspnea and anxiety, particularly in patients hospitalized for conditions like COVID-19. However, research on VR's immediate effects on exercise capacity is limited, with most studies focusing on non-immersive exergames rather than immersive VR. The potential of VR to improve exercise tolerance in patients with chronic respiratory diseases remains uncertain. Our study aims to test this hypothesis through a randomized crossover trial to assess VR's impact on dyspnea and exercise tolerance in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patient with a chronic respiratory disease requiring pulmonary rehabilitation
* Patient with dyspnea assessed as mMRC ≥ 0 (Annex 3)
* Patient undergoing pulmonary rehabilitation at the Paris Saint-Joseph Hospital
* Patient affiliated with a health insurance plan
* French-speaking patient
* Patient who has provided informed, explicit, and voluntary oral consent

Exclusion Criteria:

* Contraindications for an endurance reconditioning program (neurodegenerative diseases, severe neurological deficits, unstable cardiovascular diseases)
* History of motion sickness, vertigo, vestibular impairment, labyrinthitis
* History of seizures or other neurological or psychiatric comorbidities
* Severe visual impairments
* Patient already included in a Type 1 interventional research protocol (RIPH1)
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection
* Pregnant or breastfeeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effort duration | twice a week during up to 4 weeks
  Compare the total duration of effort during a constant-load test on a cycle ergometer between rehabilitation with VR immersion and rehabilitation alone.
  Total duration of sustained effort during a constant-load test (in seconds)."

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Paris Saint Joseph, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No